CLINICAL TRIAL: NCT05028036
Title: Personalized Lifestyle Program in Treatment Resistant Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm University (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Greger Lindberg, Clinical Professor, MD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Skandia-IBS
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized lifestyle intervention (Experimental): The intervention consists of a personalized lifestyle treatment program to address specific lifestyle issues.
  Interventions: Other: Personalized lifestyle treatment program

INTERVENTIONS:
Other: Personalized lifestyle treatment program — The personalized treatment program is based on the participants symptom profile and test results and is designed in collaboration with the participant. The treatment plan that may include several of the following components:
  * Dietary changes
  * Supplements
  * Measures to improve sleep / circadian rhythm
  * Stress management
  * Physical exercise
  The treatment plan is evaluated continuously by the participant and the therapist and adjusted accordingly. A total of 9 visits to the Nordic Clinic over one year is included in the treatment program.

SUMMARY:
Patients with treatment resistant irritable bowel syndrome (IBS) are recruited from secondary care gastroenterology clinics in Stockholm and screened for eligibility criteria. Participants follow a 12 month treatment program at Nordic Clinic, a clinic offering personalized lifestyle interventions based on the functional medicine model. In parallel with the treatment program, the participant are clinically assessed for the evaluation of the treatment after 6 months, 12 months, 18 months and 24 months

DETAILED DESCRIPTION:
Patients with treatment resistant irritable bowel syndrome (IBS) are recruited from secondary care gastroenterology clinics in Stockholm. Eligible participants are screened for eligibility criteria at a baseline visit at the Karolinska Institutet. Patients providing written informed consent for participation are invited to Nordic Clinic, a clinic offering personalized lifestyle interventions based on the functional medicine model. Before the first visit to the clinic, the participant fill out a longer questionnaire that is used for the planning of the participant's personal treatment program. At the first visit, the therapist goes through the responses together with the participant. Based on the participant's symptom profile, it is determined which tests are taken in the first step. Based on symptoms and test results, the therapist and participant come up with a treatment plan that can include several of the following components:

* Dietary changes
* Dietary supplements
* Measures to improve sleep / circadian rhythm
* Stress management
* Physical exercise
* Medicines, in exceptional cases.

The treatment plan is evaluated continuously by the participant and the therapist and adjusted accordingly.

The treatment involves a total of 9 visits to the Nordic Clinic during one year. The subsequent visits are planned by the therapist at the Nordic Clinic together with the participant.

In parallel with the treatment program, the participant makes return visits to Karolinska Institutet to collect follow-up data for the evaluation of the treatment after 6 months, 12 months, 18 months and 24 months after the start of treatment where participants are clinically assessed and fill out forms for the evaluation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fulfills Rome IV criteria for IBS
* Symptom burden on IBS-SSS >175
* No symptom relief from standard medical treatment
* No organic finding explaining the IBS symptoms (e.g. inflammation, parasites, thyroid disease, lactose intolerance, celiac disease, bile acid malabsorption)

Exclusion Criteria:

* Pregnancy
* Disease or life circumstances that prevent participation in the treatment program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2024-09-14 (Estimated); Study Completion 2025-09-14 (Estimated)

PRIMARY OUTCOMES:
Proportion recovery from diagnosis of IBS | 12 months
  Rome IV questionnaire is used to establish whether the participant fulfills the criteria for IBS at 12 months follow up

SECONDARY OUTCOMES:
Change in BS severity symptom scale score | Baseline, 6, 12, 18 and 24 months
  Assessed using the IBS severity symptom scale (IBS-SSS) which goes from 0-500. At least 150 is required to enter the study. A change of 75 is usually considered clinically relevant
Change in total symptom burden | Baseline, 6, 12, 18 and 24 months
  Assessed using Gastrointestinal symptom rating scale for IBS (GSRS-IBS) scores This scale has 13 items, each scored 1-7 so the score goes from 13-91
Change in work ability | Baseline, 6, 12, 18 and 24 months
  The participant is asked to rate its work ability and to report current employment rate and sick leave.

CONTACTS AND LOCATIONS:
Overall Officials: Greger Lindberg, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet Departmend of Medicine Hudding, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No